CLINICAL TRIAL: NCT06014450
Title: Department of Oncology, Affiliated Hospital of Guizhou Medical University Affiliated Cancer Hospital of Guizhou Medical University
Brief Title: Prophylactic Cranial Irradiation Versus Observation in Stage IV NSCLC Randomized Controlled Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guizhou Medical University (Other)
Responsible Party: Principal Investigator, Bing Lu, Chief physician, Guizhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCI for stage IV NSCLC
Record Dates: First submitted 2023-08-08; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Prophylactic Cranial Irradiation, Cumulative Incidence of Brain Metastases
Keywords: stage IV non-small cell lung cancer; PCI
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCI arm (Experimental): 72 stage IV NSCLC patients were randomly enrolled in the group. And all required to have a baseline negative MRI scan for central nervous system (CNS) disease.
  For patients with positive TKI detection, TKI combined with concurrent radiotherapy DT60-70Gy for the primary tumor. Imaging reexamination 2 months after TKI treatment confirmed the efficacy of CR, PR, and SD; meanwhile, reexamination of head MR Examination confirmed no intracranial metastasis, and PCI was performed DT 30Gy/10f.
  For patients with negative TKI detection, the treatment mode was platinum-based regimen chemotherapy combined with concurrent radiotherapy for DT60-70Gy for the primary tumor. Imaging reexamination after 2 cycles of chemotherapy confirmed the efficacy of CR, PR, and SD, and skull MR Examination confirmed that there was no intracranial metastasis. PCI DT: 30Gy/10f.Systematic imaging examinations in the first month following systemic treatment, every 3 months in 2 years, and every 6 months in 5 years.
  Interventions: Radiation: Prophylactic Cranial Irradiation for experiment arm
- observation arm (Placebo Comparator): 72 stage IV NSCLC enrolled in the observation group. And all required to have a baseline negative magnetic resonance imaging (MRI) scan for central nervous system (CNS) disease. For patients with positive TKI detection, TKI combined with concurrent radiotherapy DT60-70Gy for the primary tumor.
  For patients with negative TKI detection, the treatment mode was platinum-based regimen chemotherapy combined with concurrent radiotherapy for DT60-70Gy for the primary tumor. Imaging reexamination after 2 cycles of chemotherapy confirmed the efficacy of CR, PR, and SD, and skull MR Examination confirmed that there was no intracranial metastasis. then observation. Systematic imaging examinations in the first month following systemic treatment, every 3 months in 2 years, and every 6 months in 5 years.
  Interventions: Radiation: Prophylactic Cranial Irradiation for experiment arm

INTERVENTIONS:
Radiation: Prophylactic Cranial Irradiation for experiment arm — Prophylactic Cranial Irradiation DT30Gy/10f

SUMMARY:
Lung cancer has remained the leading cause of cancer-related deaths worldwide. An important and frequent cause of morbidity in this patient group is the development of brain metastases (BM). Lung cancer represents the leading cause of BM, and previous reports have shown that approximately 40% of patients will develop BM throughout their disease. Additionally, due to the improved use of advanced imaging techniques as part of routine initial staging. Another factor to consider is the considerably prolonged survival in patients with lung cancer as a direct result of the medical advances that have improved systemic disease control in the past 2 decades.

The development of BM has recognized as one of the most detrimental factors for patient prognosis, with a negative impact on quality of life (QoL), concomitant neurocognitive disorders, and, importantly, a significant decrease in OS.

RTOG 0214 shows that In patients with stage III disease without progression of disease after therapy, PCI decreased the rate of BM. NVALT-11/DLCRG-02 Study shows that PCI significantly decreased the proportion of patients who developed symptomatic brain metastases with an increase in low-grade toxicity. In conclusion, PCI improved DFS and decreased the risk of BM in patients with LA-NSCLC.Recent studies suggest NSCLC, including stage IV NSCLC, PCI significantly decreased CBM in addition to increasing progression-free survival and OS.

At present, few studies on whether prophylactic radiation therapy can reduce the rate of brain metastasis and OS in stage IV NSCLC. In this randomized controlled study of stage IV NSCLC, we investigated whether PCI reduces the chance of brain metastases and whether it has a survival benefit.

DETAILED DESCRIPTION:
Group sample sizes of 72 in Group 1 and 72 in Group 2 achieve 90.140% power to detect a difference between the group proportions of 0.3100. The Group 2 proportion is 0.0700. The Group 1 proportion is assumed to be 0.1700 under the null hypothesis and 0.3800 under the alternative hypothesis. The test statistic used is the one-sided Z test (unpooled). The significance level of the test is 0.0250.

For all patients with positive TKI detection, TKI combined with concurrent radiotherapy DT60-70Gy for the primary tumor. Imaging reexamination 2 months after TKI treatment confirmed the efficacy of CR, PR, and SD; meanwhile, reexamination of head MR Examination confirmed no intracranial metastasis.

For all patients with negative TKI detection, the treatment mode was platinum-based regimen chemotherapy combined with concurrent radiotherapy for DT60-70Gy for the primary tumor. Imaging reexamination after 2 cycles of chemotherapy confirmed the efficacy of CR, PR, and SD, and skull MR Examination confirmed that there was no intracranial metastasis.

Then,for the experiment arm,patients will receive prophylactic cranial irradiation DT: 30Gy/10f. Followed systematic imaging examinations in the first month following systemic treatment, every 3 months in 2 years, and every 6 months in 5 years.

For the observation arm,without prophylactic cranial irradiation,Followed systematic imaging examinations in the first month following systemic treatment, every 3 months in 2 years, and every 6 months in 5 years.

The primary end point was incidence of brain metastases（CBM）, PFS, and the secondary end point was OS、quality of life (QoL), concomitant neurocognitive disorders。

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically or cytologically confirmed NSCLC; patients with clinical stage IV and no brain metastases [AJCC 8th edition]; no previous treatment
* Age 18 ~ 80 years old, body condition score ECOG 0 ~ 2 or KPS≥70;
* No contraindications such as radiotherapy, EGFR-TKI, chemotherapy, or immunotherapy;
* IMRT is required for primary tumor radiotherapy. DT: 60-70Gy
* Metastases are treated with three-dimensional radiotherapy (IMRT/SRT/SBRT/VMAT, etc.) and large segmentation radiotherapy.
* The subject must have no major organ dysfunction or laboratory tests that meet the following requirements:
* Hematological tests such as liver and kidney function were in the normal range of laboratory standards;
* Cardiac function: electrocardiogram excluded organic arrhythmia;
* Pulmonary function test: FEV1>50%, mild-moderate lung function limited.
* Signed informed consent before treatment (radiotherapy, chemotherapy, immunization, targeted drug therapy); The patient had good compliance with the treatment and follow-up received.

Exclusion Criteria:

* Patients with brain metastasis;
* Stage IV NSCLC patients with malignant pleural effusion, pericardial effusion and other serous effusion;
* Patients with extensive liver metastasis and intrapulmonary metastasis that have seriously affected liver and lung function;
* Patients with uncontrolled hypertension, diabetes, unstable angina, history of myocardial infarction, or symptomatic congestive heart failure or uncontrolled arrhythmia within the past 12 months; Have a clinically clear diagnosis of heart valve disease; The disease active phase of bacterial, fungal, or viral infection; Mental disorders; Severe impaired lung function;
* Pregnant or lactating patients;
* Patients with a history of active malignancy other than small cell lung cancer prior to enrollment; Non-melanoma skin basal cell carcinoma, in situ cervical cancer, cured early prostate cancer excepted;
* Patients with an allergy and known or suspected allergy to any investigational drug for which no alternative medicine is available;
* Patients with poor compliance;
* Researchers consider it inappropriate to participate in this experiment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
PFS is defined as the duration of time from start of treatment to time of progression or death,whichever occurs first.,CBM is defined as cumulative incidence of brain metastases. | Systematic imaging examinations in the first month following systemic treatment, every 3 months in 2 years, and every 6 months in 5 years.

SECONDARY OUTCOMES:
Overall survival is defined as the time interval from date of diagnosis to date of death from any cause. Quality of life and neurocognitive function. | Systematic imaging examinations in the first month following systemic treatment, every 3 months in 2 years, and every 6 months in 5 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Guizhou Cancer Hospital, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: No